CLINICAL TRIAL: NCT01058889
Title: Tele-Diab: Electronic Diary for Patients With Type 2 Diabetes Mellitus
Acronym: Tele-Diab
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Bernhard Ludvik, MD, Prof., Medical University Vienna,
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 352/2006
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus Type 2; Insulin Resistance
Keywords: Diabetes mellitus Type 2; Telemedicine; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedical device (Experimental): Patient will receive a blood glucose measurement device and a telemedical device to monitor blood glucose measurements.
  Interventions: Device: Telemedical device
- Treatment as usual (No Intervention)
  Interventions: Device: Telemedical device

INTERVENTIONS:
Device: Telemedical device — Monitoring of blood glucose,insulin dose, blood pressure, lifestyle factors with the telemedical device. Monitoring of system availability, percentage of data transfer, acceptance.
  Other Names: mobile phone

SUMMARY:
The purpose of the study is to show if telemonitoring and automated feedback regarding glucose management, physical activity, blood pressure, and body weight improves treatment of patients with insulin dependent Type 2 Diabetes mellitus.

DETAILED DESCRIPTION:
In this clinical trial 50 patients with insulin dependent type 2 diabetes will be randomised in two study arms: monitoring of blood glucose and blood pressure using a telemedical device or in an arm with treatment as usual. Patients will the following measurement devices: blood glucose, blood pressure. Both devices can communicate with a mobile phone, which will also be provided to the patients. The mobile phone will transfer the data to a central, safe server. Patients will receive automated reminder/feedback. Caregivers can evaluate the transferred data whenever necessary via a web-based access. Data will be presented in tables as well as trend figures.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 2, age 18-70 years, able to use a mobile phone

Exclusion Criteria:

* Pacemaker, intracardial defibrillator, no cure planned within the active study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
System availability, acceptance, transmission rate | 3 months

SECONDARY OUTCOMES:
HbA1c | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Ludvik, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Allgemeines Krankenhaus, Vienna, Austria